CLINICAL TRIAL: NCT01484106
Title: Cardiac Output Monitoring Managing Intravenous Therapy (COMMIT) to Treat Emergency Department Severe Sepsis
Acronym: COMMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheetah Medical Inc. (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01-CM-2011
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): Patients will be randomized (1:1, stratified by site, in permutation blocks of 4) to the "Treatment" or "Standard Care" arms.
  Interventions: Other: Fluid Resuscitation
- Control (Active Comparator): Standard of Care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Fluid Resuscitation — In the Treatment group, this information will be used in a specific 4-hour treatment algorithm to guide fluid administration that is summarized in Figure 1. The information provided by the NICOM in response to the fluid bolus will be used to assess whether the subject is "fluid responsive" (FR).
  Arms: Treatment group
Other: Standard of Care — Standard of Care
  Arms: Control

SUMMARY:
The primary objective of this study is to test whether a fluid resuscitation protocol guided by non-invasive hemodynamic measures reduces the progression of organ dysfunction (defined by an increase in the Serial Organ Failure Assessment Score ≥ 1 over the first 72 hours) in sepsis patients presenting to the Emergency Department without evidence of shock.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients > 18 years with old suspected or confirmed infection
2. At least two of the following four criteria (SIRS):

   1. Temperature > 38 or < 36o C
   2. Heart rate > 90 bpm
   3. Respiratory rate > 20 bpm or PaCO2< 32 mmHg
   4. White blood cell count >12,000 or <4,000 per mm3; or >10% bandemia
3. Lactate ≥2.0 and ≤4.0 mMol/L
4. Enrollment within 6 hours of ED presentation within 2.5 hours of meeting eligibility criteria

Exclusion Criteria:

1. Age < 18 years
2. On vasopressor therapy
3. Systolic blood pressure < 90 mmHg
4. Received more than 3-liter crystalloid fluid prior to randomization
5. Patient presenting with pulmonary edema
6. Patient presenting with acute coronary syndrome
7. Patient presenting with new onset cardiac arrhythmia
8. Patient presenting with trauma, including burns
9. Patient requires immediate surgery
10. Patient presenting with stroke
11. Patient with end stage renal disease on renal replacement therapy
12. Patient with known pregnancy
13. Patient being treated with immunosuppressive therapy for organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
sequential organ failure assessment score increases by greater or equal to 1 point from the baseline score within 72 hours of study enrollment. | 72 hours
  A patient will be considered to have progressive organ dysfunction if their "Sequential Organ Failure Assessment" (SOFA) score increases by ≥1 point from their baseline score within 72 hours of study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Nate Shapiro, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (12):
- United States (12):
  - University of Alabama, Birmingham, Alabama
  - University of California, Sacramento, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Northwester University, Evanston, Illinois
  - MGH, Boston, Massachusetts
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Dr. Nate Shapiro, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NY Methodist Hospital, Brooklyn, New York
  - Humility of Mary Health Partners, Youngstown, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Sentara Norfolk General Hospital, Norfolk, Virginia